CLINICAL TRIAL: NCT06511102
Title: A Randomized Controlled Trial on the Impact of Using Generative Artificial Intelligence on Analytical Writing Performance and Cognitive Abilities
Brief Title: Impact of GPT Use on Essay Writing Performance and Cognitive Abilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Simiao Chen, Professor, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: S-117/2024
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Cognitive Change; Well-Being, Psychological
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): In the intervention arm, participants are instructed to use ChatGPT for assistance to complete an analytical writing task.
  Interventions: Behavioral: GPT Support
- Control arm (No Intervention): In the control arm, participants are instructed to complete an analytical writing task independently without access to any technology assistance.

INTERVENTIONS:
Behavioral: GPT Support — The computer interface used for the essay writing task follows a split-screen design. The writing instructions and text input field are administered on a survey platform, placed on the left half of the screen. ChatGPT is placed on the right half of the screen for technology assistance.
  Arms: Intervention arm

SUMMARY:
The goal of this randomized controlled lab experiment is to examine if using generated artificial intelligence (AI) technology will affect people's academic performance and cognitive abilities in the context of analytical writing among college students. The main questions it aims to answer are:

1. Does using the technology affect students' writing performance?
2. Does using the technology affect students' cognitive effort during the writing process?

Participants will be randomly assigned to either a control group, which is writing without AI assistance, or an experimental group, which is writing with the assistance of ChatGPT. Researchers will compare the two groups to see if ChatGPT affects students' writing performance and cognitive effort.

For each participant, the lab experiment will last for no more than 1.5 hours. An eye-tracker will monitor the participant's gaze activities and pupil size. A functional near-infrared spectroscopy (fNIRS) will monitor the participant's brain activities in the frontal lobe. During the experiment, participants will be asked to:

1. Read learning materials on analytical writing techniques.
2. Based on the previously provided materials, complete an analytical writing assignment that will take approximately 30 minutes either with or without the aid of ChatGPT.
3. Answer survey questions about their experience with the writing assignment, attitudes on using ChatGPT, and demographic backgrounds.

ELIGIBILITY:
Inclusion Criteria:

* Full-time university student.
* Able to read and write in English.
* Use the computer most days of the week.
* Have not taken, nor currently preparing for, the Graduate Record Examinations (GRE).
* Do not wear glasses (contact lenses are allowed).
* Have no eye impairment.
* Not currently taking any opioids, epinephrine, or anti-hypertensive drugs.
* During the experiment, not wearing any makeup around the eyes.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Writing Performance | 1.5 hours
  The essay writing task is derived from the Analytical Writing section in the Graduate Record Examinations (GRE), which is a worldwide and standardized computer-based exam developed by the Educational Testing Service (ETS). The participants' essays will be scored on a scale from 0 to 6 by an automatic and validated third-party scoring tool that is also developed by ETS.
Cognitive Effort Measured by Pupil Size | 1.5 hours
  Cognitive effort is quantified by monitoring changes in pupil size. To achieve this, pupil diameters are recorded throughout the writing task using a near-infrared eye tracker, specifically the Tobii Pro Fusion model. At the start of the experiment, individual baseline pupil diameters are measured during a 30-second relaxation task.

SECONDARY OUTCOMES:
Self-Perception of Writing Performance | 1.5 hours
  This is a one-item scale:
  Using the same grading rubric from before, what score do you think your essay should get (0 being the lowest and 6 being the highest)?
  The score ranges from 0 to 6. A higher score indicates higher self-perceived writing performance. The variable is treated as a continuous variable.
Self-Perception of Cognitive Effort | 1.5 hours
  This is a one-item Likert scale adapted from the National Aeronautics and Space Administration-task load index (NASA-TLX; Hart, 2006; Hart & Staveland, 1988):
  On a scale of 1 to 7, rate how hard you have to work to accomplish your level of performance.
  The Likert score ranges from 1 to 7 (1 being "very low" and 7 being "very high"). A higher score indicates higher self-perceived cognitive effort. The variable is treated as a continuous variable.
  References:
  1. Hart, S. G. (2006). Nasa-Task Load Index (NASA-TLX); 20 Years Later. Proceedings of the Human Factors and Ergonomics Society Annual Meeting. https://doi.org/10.1177/154193120605000909
  2. Hart, S. G., & Staveland, L. E. (1988). Development of NASA-TLX (Task Load Index): Results of empirical and theoretical research. In Advances in Psychology (Vol. 52, pp. 139-183). North-Holland.
Cognitive Effort Measured by Cortical Hemodynamic Activity in the Frontal Lobe | 1.5 hours
  Cognitive Effort is quantified by monitoring changes in the cortical hemodynamic activity in the frontal lobe. To achieve this, the brain activity is recorded throughout the writing task using a functional near-infrared spectroscopy (fNIRS), specifically the NIRSport2 model.
Self-Perception of Stress | 1.5 hours
  This is a one-item Likert sub-scale adapted from the Primary Appraisal Secondary Appraisal scale (PASA; Gaab, 2009; Pollak et al., 2020):
  On a scale of 1 to 7, how much would you agree or disagree with the following statement on perceived stress: The analytical writing assignment was stressful to me.
  The Likert score ranges from 1 to 7 (1 being "strongly disagree" and 7 being "strongly agree"). A higher score indicates higher self-perceived stress. The variable is treated as a continuous variable.
  References:
  1. Gaab, J. (2009). PASA-Primary Appraisal Secondary Appraisal. A questionnaire for the assessment of cognitive appraisals of situations. Verhaltenstherapie, 19(2), 114-115.
  2. Pollak, A., Paliga, M., Pulopulos, M. M., Kozusznik, B., & Kozusznik, M. W. (2020). Stress in manual and autonomous modes of collaboration with a cobot. Computers in Human Behavior, 112, 106469. https://doi.org/10.1016/j.chb.2020.106469
Self-Perception of Challenge | 1.5 hours
  This is a one-item Likert sub-scale adapted from the Primary Appraisal Secondary Appraisal scale (PASA; Gaab, 2009; Pollak et al., 2020):
  On a scale of 1 to 7, how much would you agree or disagree with the following statement on perceived challenge: I find the analytical writing assignment a challenge.
  The Likert score ranges from 1 to 7 (1 being "strongly disagree" and 7 being "strongly agree"). A higher score indicates higher self-perceived challenge. The variable is treated as a continuous variable.
  References:
  1. Gaab, J. (2009). PASA-Primary Appraisal Secondary Appraisal. A questionnaire for the assessment of cognitive appraisals of situations. Verhaltenstherapie, 19(2), 114-115.
  2. Pollak, A., Paliga, M., Pulopulos, M. M., Kozusznik, B., & Kozusznik, M. W. (2020). Stress in manual and autonomous modes of collaboration with a cobot. Computers in Human Behavior, 112, 106469. https://doi.org/10.1016/j.chb.2020.106469
Self-Efficacy in Writing | 1.5 hours
  This is a sixteen-item Likert scale that measures three dimensions of writing self-efficacy: ideation, convention and self-regulation (Bruning et al., 2013). The Likert score ranges from 1 to 7 (1 being "strongly disagree" and 7 being "strongly agree"). A higher score indicates higher self-efficacy. The three dimensions will be treated separately, each as a continuous variable.
  Reference:
  1. Bruning, R., Dempsey, M., Kauffman, D. F., McKim, C., & Zumbrunn, S. (2013). Examining dimensions of self-efficacy for writing. Journal of educational psychology, 105(1), 25.
Situational Interest in Analytical Writing | 1.5 hours
  This is a four-item Likert scale adapted from the situational interest scale (Hulleman et al., 2010). This scale measures participants' situational interest in analytical writing:
  On a scale of 1 to 7, how much would you agree or disagree with the following statements on your interest in the analytical writing assignment that you just completed?
  1. The analytical writing assignment was interesting.
  2. Working on the essay was fun.
  3. I enjoyed writing the essay.
  4. The analytical writing assignment was enjoyable.
  The Likert score ranges from 1 to 7 (1 being "strongly disagree" and 7 being "strongly agree"). A higher score indicates higher situational interest. The variable is treated as a continuous variable.
  Reference:
  1. Hulleman, C. S., Godes, O., Hendricks, B. L., & Harackiewicz, J. M. (2010). Enhancing interest and performance with a utility value intervention. Journal of Educational Psychology, 102(4), 880.
Behavioral Intention in Using ChatGPT | 1.5 hours
  This is a two-item Likert scale that measures participants' behavioral intention in using ChatGPT in the future for essay writing tasks (Albayati, 2024):
  On a scale of 1 to 7, how much would you agree or disagree with the following statements on using ChatGPT in essay writing assignments?
  1. If I have access to ChatGPT, I would use it for essay writing tasks.
  2. I plan to use ChatGPT in the future if I have an essay writing task.
  The Likert score ranges from 1 to 7 (1 being "strongly disagree" and 7 being "strongly agree"). A higher score indicates higher behavioral intention in using ChatGPT. The variable is treated as a continuous variable.
  Reference:
  1. Albayati, H. (2024). Investigating undergraduate students' perceptions and awareness of using ChatGPT as a regular assistance tool: A user acceptance perspective study. Computers and Education: Artificial Intelligence, 6, 100203. https://doi.org/10.1016/j.caeai.2024.100203

CONTACTS AND LOCATIONS:
Overall Officials: Till Bärnighausen, Principal Investigator — Heidelberg Institute of Global Health
Locations (1):
- Core Facility for Neuroscience of Self-Regulation, Heidelberg University, Heidelberg, Germany

REFERENCES:
- [Derived] Chen Y, Wang Y, Wustenberg T, Kizilcec RF, Fan Y, Li Y, Lu B, Yuan M, Zhang J, Zhang Z, Geldsetzer P, Chen S, Barnighausen T. Effects of generative artificial intelligence on cognitive effort and task performance: study protocol for a randomized controlled experiment among college students. Trials. 2025 Jul 11;26(1):244. doi: 10.1186/s13063-025-08950-3. PMID 40646586